CLINICAL TRIAL: NCT00360321
Title: Descriptive Study of a French Sample of "at Risk" and Pathological Gamblers Followed in a French Structure Specialised in Addictive Disorders.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Other Study IDs: BRD 06/5-M
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-07

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
International surveys about pathological gambling estimate that there are about 1 to 3 per cent of gamblers who develop a pathological behavior about gamble.In France, pathological gambling is not a priority of public health, in contrast with other addictive disorders, like alcoholism or nicotine addiction. The aim of our study is to describe accurately for the first time in France, a sample of "at risk" and pathological French gamblers. We want to collect socio-demographical and clinical data from this subjects (story of the addictive behaviour, co morbidities, and more specifically, detailed study of pathological gamblers' personality), in order to compare our data with those of international literature.Secondarily, we want to test the feasibility of this kind of detailed evaluations for another study planned for 2007-2008 and which purpose will be to compare pathological gamblers' personality characteristics according to the kind of game that they mainly practice.The participation at the study will be proposed to every patient consulting in the "service d'addictologie du CHU de Nantes". The study consists in a single evaluation (about 8 hours) with standardized tools used all other the world.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70
* Consulting or ex-consulting since 2000 in the "service d'addictologie du CHU de Nantes"
* Who meet sufficient criteria of pathological or "at risk" gambling in the DSM-IV section about pathological gambling
* Who accept to participate
* Who give their consent
* Who don't have any exclusion criteria

Exclusion Criteria:

* Gambling behaviour directly and chronologically explain by an acute maniac fit
* Superior function trouble
* Who don't agree to participate
* Difficulties in reading or writing in French

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Venisse Jean Luc, Professor, Principal Investigator — Nantes University Hospital